CLINICAL TRIAL: NCT02498717
Title: Preliminary Efficacy and Cost-effectiveness Analysis of a Cold and Active Intermittent Compression Therapy Technique for Traumatic Calcaneus or Ankle Fractures
Brief Title: Preliminary Review of Cold and Active Compression Therapy for Traumatic Calcaneus or Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Cool Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 539147
Record Dates: First submitted 2015-03-31; First posted 2015-07-15 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RICE (control) (Active Comparator): Standard of Care procedures including ice and elevation.
  Interventions: Other: RICE
- Cryocompression (experimental) (Experimental): treatment using the GameReady cryotherapy system
  Interventions: Device: GameReady

INTERVENTIONS:
Device: GameReady — Cryotherapy and compression
  Arms: Cryocompression (experimental)
Other: RICE — SOC ice and elevation
  Arms: RICE (control)

SUMMARY:
This study will examine the initial efficacy and cost-effectiveness of using the cryocompression therapy model both pre-operatively and post-operatively in patients that have recently suffered a traumatic calcaneus or ankle fracture compared to the standard pre-operative RICE therapy procedures.

DETAILED DESCRIPTION:
Initial research has shown that cryocompression therapy applied post-operatively has been effective in reducing recovery time and improving health and pain factors related to patient recovery. However, there has been limited research into how this translates into positive economic outcomes for both the hospital and the patient. In addition, it can be reasonably hypothesized that the use of the cryocompression therapy system before surgery will lead to an increased rate of reduction in swelling necessary to allow proper operative procedures to take place when compared to the standard ice and elevation (RICE) therapy techniques and cryocompression therapy applied only post-operatively. This should lead to decreased hospital costs and possible improved patient outcomes related to recovery.

Study Objectives This study will examine the initial efficacy and cost-effectiveness of using the cryocompression therapy model both pre-operatively and post-operatively in patients that have recently suffered a traumatic calcaneus or ankle fracture compared to the standard pre-operative RICE therapy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Able to provide informed consent
3. Recent calcaneus or ankle fracture requiring fixation
4. Injury is determined (by physician) to be an isolated, closed, low-energy bimalleolar fracture

Exclusion Criteria:

1. Unable to provide informed consent
2. History of Dementia or mental instability
3. No recent additional fractures (within one year) at or around injury site
4. Persons with symptoms of any kind of psychosocial disorder
5. Any condition that the clinician feels would contraindicate for the postoperative test or control treatments
6. Any conditions that would contraindicate using the Game Ready
7. If the patient is prevented from transfer to the OR due to reasons other than medically necessary

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Time until surgery/Time until discharge (LOS) | Measured from intake to time of surgery (days) and upon discharge from hospital (days). Estimated period of time to be up to 10 days until surgery and up to 7 days after surgery until discharge.
  Reduction in length of stay (LOS) and time of effect (pre-/post-op)
Change in Swelling as measured by point of largest swollen area (tape measure) | Measured at baseline and all follow-up assessments (2, 8, 16, & 24-weeks post-op)
  Measured at circumference of swelling point
Total Narcotic Use as recorded on MR chart and Knee Pain Assessment | Measured daily while inpatient (approx 2-3 days) and retroactively at all follow-up assessments (2, 8, 16, & 24-weeks post-op)
  reported as yes/no and amount/type on assessment form
Change in Patient reported pain as measured on VAS and Knee Pain Assessment | Reported at baseline, daily while inpatient (approx 2-3 days), and at all follow-up assessments (2, 8, 16, & 24-weeks post-op)
  As reported by VAS scale

SECONDARY OUTCOMES:
Change in Quality of Life (QALY) as measured on QOL and SF-8 | At baseline and all follow-up assessments (2, 8, 16, & 24-weeks post-op)
  Quality of Life by QALY score

CONTACTS AND LOCATIONS:
Overall Officials: Brian Vickaryous, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States